CLINICAL TRIAL: NCT05970263
Title: IKANOS: A Prospective, Open-Label, Minimally Interventional Hybrid Study in the US Comparing Initiation of Breztri Maintenance Versus Any Non-Triple Inhaled Therapy at Discharge After a Hospitalization for a COPD Exacerbation
Brief Title: IKANOS: Breztri Maintenance Versus Any Non-Triple Inhaled Therapy After Hospitalization for a COPD Exacerbation in the US
Acronym: IKANOS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry); Premier Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5980C00034
Record Dates: First submitted 2023-06-27; First posted 2023-08-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: COPD
Keywords: COPD;; readmissions;; maintenance therapy;; triple therapy;; real-world evidence;; hospital discharge;; mortality;; cardiopulmonary events,; exacerbations
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Glycopyrrolate; Formoterol Fumarate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Breztri (Experimental): 1. Interventional Arm: patients receive :
  1. First dose of Breztri during hospitalization and discharge with 7-day Breztri inhaler
  2. Breztri refills to cover 12-month follow-up period, mailed in 90-day supply from a central pharmacy. Emergency resupply is also available if needed.
  Interventions: Drug: Budesonide/glycopyrrolate/formoterol fumarate (Breztri Aerosphere) 320 μg/18 μg/9.6 μg administered as two inhalations, twice daily.
- External Comparator - Non-Triple (Other): 2. External Comparator Arm: patient who receive any non-triple inhaled therapy following a hospitalization for severe COPD exacerbation. This arm will be constructed of de-Identified patient.
  Interventions: Other: External Comparator

INTERVENTIONS:
Drug: Budesonide/glycopyrrolate/formoterol fumarate (Breztri Aerosphere) 320 μg/18 μg/9.6 μg administered as two inhalations, twice daily. — 2 inhalations twice daily administered by oral inhalation, from a metered dose inhaler, over a 12-month follow-up period.
  Arms: Breztri
Other: External Comparator — Received any inhaled therapy, excluding triple inhaled maintenance therapy, during index hospitalization and refilled within 30 days before or after discharge from index hospitalization
  Arms: External Comparator - Non-Triple

SUMMARY:
This study will evaluate whether prompt initiation and maintenance of Breztri (a triple therapy) following a severe COPD exacerbation hospitalization, is associated with a lower risk of all-cause readmissions at 90 days post-discharge, compared to receiving any non-triple inhaled therapy.

DETAILED DESCRIPTION:
IKANOS is a prospective, open-label, minimally interventional Hybrid Study in the US Comparing Initiation of Breztri Maintenance versus Any Non-Triple Inhaled Therapy at Discharge after a Hospitalization for a COPD Exacerbation.

The interventional arm will be comprised of around 1000 patients for whom Breztri maintenance is prescribed, and the first dose is received prior to hospital discharge (the "index discharge") after a severe COPD exacerbation (the index admission).

At the end of the recruitment period of the interventional arm, the external comparator arm will be constructed from real-world data of patients contemporaneous with those in the interventional arm, from the same or similar integrated delivery network as the interventional arm and who are similar in key clinical and demographic characteristics.

Patients will be followed-up through their data and call center contact for up to 12 months.

ELIGIBILITY:
Patients are included into the study if they meet the following criteria :

1. Adults aged 40 years and above as of the index hospitalization admission date (for the intervention arm only).
2. Primary or secondary diagnosis of COPD as documented in the database on or before admission.
3. Hospital admission for a COPD exacerbation (primary or secondary cause) (ie, the index admission).
4. Availability of at least 6 months of data in the PHD-LRx-Dx database prior to the index admission (for the comparator arm only).
5. Additional inclusion criteria for the interventional arm:

   1. Willingness to use Breztri as an inhaled maintenance medication as prescribed by their physician.
   2. Willingness and ability to sign informed consent during index admission and before discharge.
   3. Availability of home-based access to telephone calls.
   4. Availability of home-based access to the internet for PRO measurement and inhaler training materials.
   5. Willingness to be contacted by a qualified medical professional for safety monitoring.
   6. Willingness and ability to participate, on their own or through the assistance of their caregivers, in remote, online patient-reported outcome measurement at designated intervals
   7. Physician decision that patient is eligible for treatment with Breztri according to the approved USPI.
   8. Any females of childbearing potential must be using a form of highly effective methods of contraception and have a negative urine pregnancy test result
6. Additional inclusion criterion for the comparator arm:

   1. Received non-triple inhaled therapy for COPD within 30 days prior to discharge or up to 30 days post-discharge, including:

      * ICS/LABA.
      * LABA/LAMA.
      * ICS.
      * LABA.
      * LAMA.
      * SABA/SAMA.
      * SABA.
      * SAMA.
      * Other inhaled COPD therapy not classified as triple therapy.

Exclusion Criteria:

Patients are excluded from the study if they meet any of the following criteria:

1. Having received triple inhaled maintenance therapy (fixed-dose, or open) for COPD or other indications 6 months prior to index admission.
2. Any documented use of respiratory biologics 6 months prior to index admission.
3. Patients on palliative care, including hospice.
4. Discharge to institutional care other than a rehabilitation facility (eg, other hospital, or similar). Patients discharged to rehabilitation facility are eligible to participate. Note: Because patients are enrolled in the intervention arm prior to discharge, this criterion should be assessed using the working knowledge of the treating physician at the time of patient enrollment.
5. Mortality on or before index discharge.
6. Conditions including lung surgery (excluding thoracentesis or chest tube insertion or thoracostomy) in 6 months prior to index admission, history of pulmonary lobectomy, cystic fibrosis, interstitial lung disease, lung cancer, or alpha-1 antitrypsin deficiency (A1ATD) inducing severe disease as recorded in the PHD-LRx-Dx database.
7. For females only - currently pregnant (confirmed with positive pregnancy test) or breast-feeding or planning to become pregnant in the year following index discharge.
8. Additional exclusion criteria for the interventional arm:

   1. Discharged on a triple inhaled maintenance therapy in addition to Breztri.
   2. Patients who have a history of hypersensitivity to β2-agonists, budesonide or any other corticosteroid components, glycopyrronium or other muscarinicanticholinergics, or any component of the MDI.
   3. Patients who are clinically unstable, ie, still admitted within the intensive care unit,with ongoing dyspnea, requiring vasopressors or round-the-clock positive airway pressure ventilatory support.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-19 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with an all-cause readmission | 90 days post-index discharge

SECONDARY OUTCOMES:
Number of all-cause readmissions | 90 days post-index discharge
Time to first all-cause readmission | 1 year post-index discharge
Proportion of patients with all-cause readmissions | 30 days and 1 year post-index discharge
number of all-cause readmissions per time period | 30 days and 1 year post-index discharge
proportion of patients experiencing COPD moderate/severe exacerbations | 30 days, 90 days and 1 year post-index discharge
proportion of patients experiencing COPD severe exacerbations | 30 days, 90 days, and 1 year post-index discharge
number of COPD moderate/severe exacerbations per time period | 30 days, 90 days, and 1 year post-index discharge
number of COPD severe exacerbations per time period | 30 days, 90 days, and 1 year post-index discharge
time to first COPD moderate/severe exacerbations | 1 year post-index discharge
time to first COPD severe exacerbations | 1 year post-index discharge
proportion of patients experiencing all-cause mortality | 90 days and 1 year post-index discharge
time to all-cause mortality | 1 year post-index discharge

CONTACTS AND LOCATIONS:
Overall Officials: Igor Barjaktarevic, MD, PhD, Principal Investigator — David Geffen School of Medicine

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at
URL: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.